CLINICAL TRIAL: NCT03031015
Title: Randomized Comparison of Cemented K-wire Fixation and Plating of Shaft Fractures of Proximal Phalanges
Brief Title: Cemented K-wire Fixation vs Plating for Finger Fractures
Acronym: CKFPFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THHMU201701
Record Dates: First submitted 2017-01-19; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Closed Fracture of Finger; Finger Fracture Open
Keywords: Reduction, Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Electroplating

STUDY DESIGN:
Intervention Model Description: Patients with proximal phalangeal fractures of fingers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cemented K-wire Fixation (Experimental): The mean age of group A was 41 years (range, 18-63 years). There were 56 male and 11 female patients. The mean time from injury to operation was 5±4.53 days. Injured digits included index (n=24), long (n=19), ring (n=9), and little (n=15) fingers. Types of fractures were transversal (n=31), oblique or spiral (n=14), and comminuted (n=22) fractures. The patients were treated with Cemented K-wire Fixation.
  Interventions: Device: Cemented K-wire Fixation; Device: Plating
- Plating (Active Comparator): The mean age of group A was 39 years (range, 19-61 years). There were 51 male and 13 female patients. The mean time from injury to operation was 6±5.53 days. Injured digits included index (n=21), long (n=17), ring (n=10), and little (n=16) fingers. Types of fractures were transversal (n=34), oblique or spiral (n=11), and comminuted (n=19) fractures.The patients were treated with Plating.
  Interventions: Device: Cemented K-wire Fixation; Device: Plating

INTERVENTIONS:
Device: Cemented K-wire Fixation — Fractures were reduced and then fixed with cemented K-wires.
Device: Plating — Fractures were reduced and then fixed with Plate.

SUMMARY:
To introduce a novel external-fixation technique using the combination of K-wires and cement. For comparison, we also included another group of patients who were treated using a mini plate and screw system. Bone healing, range of motion of the fingers, costs of treatments, and patient satisfaction were assessed.

DETAILED DESCRIPTION:
Shaft fractures of the proximal phalanx are common injuries that may significantly affect hand function. Good fracture stability to allow early mobilization of joints and thus early return of function. The objective of this report is to introduce a novel external-fixation technique using the combination of K-wires and cement. For comparison, we also included another group of patients who were treated using a mini plate and screw system. A total of 104 patients (131 fingers) were randomly allocated into group A (56 patients) and B (51 patients). Patients in group A were treated with cemented K-wire fixation; and patients in group B were treated with conventional mini-plate. Bone healing, range of motion of the fingers, costs of treatments, and patient satisfaction were assessed.

ELIGIBILITY:
Inclusion Criteria:

* patient aged between 18 and 65 years;
* acute fractures within 15 days;
* closed fracture or open injury with small wound less than 1.5 cm;
* involvement of proximal phalanges of index to little fingers; shaft fractures;
* at least 5 mm in length of the most distal and proximal fragments so that the K-wires or screws can be engaged;
* oblique, spiral, and comminuted fractures;
* normal opposite hand for comparison.

Exclusion Criteria:

* patients younger than 18 years are excluded because of skeletal immaturity;
* patients older than 65 years are excluded because of possible osteoporosis;
* severe open injury or crush injuries; tendon or neurovascular injuries; - involvement of articular surface;
* old fractures exceeding 15 days because close reduction was most likely difficult;
* a combined tendon, nerve, or artery injuries or diseases; diabetes, gout, ganglion;
* osseous tumors, and other disease affecting bony structures and joint motion;
* patients who declined to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2014-05-01 (Actual)

PRIMARY OUTCOMES:
Bone healing | Up to 12 weeks. From date of randomization until the date of first documented progression from any cause, which is assessed up to 12 weeks.
  Time of bone healing.

SECONDARY OUTCOMES:
Joint motion | Up to 2 years. From date of randomization until the date of second documented progression from any cause, which is assessed up to 2 years.
  Range of motion of MCP, PIP, and DIP joints.

OTHER OUTCOMES:
Patient satisfaction. | Up to 2 years. From date of randomization until the date of third documented progression from any cause, which is assessed up to 2 years.
  Patient self assessment based on 100-mm visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, MD, Study Chair — Third Hospital of Hebei Medical University; Xinzhong Shao, MD, Principal Investigator — Third Hospital of Hebei Medical University
Locations (1):
- Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No
No plan to share the IPD data.

REFERENCES:
- [Result] Miller L, Ada L, Crosbie J, Wajon A. Pattern of recovery after open reduction and internal fixation of proximal phalangeal fractures in the finger: a prospective longitudinal study. J Hand Surg Eur Vol. 2017 Feb;42(2):137-143. doi: 10.1177/1753193416670591. Epub 2016 Oct 4. PMID 27702779
- [Result] Borbas P, Dreu M, Poggetti A, Calcagni M, Giesen T. Treatment of proximal phalangeal fractures with an antegrade intramedullary screw: a cadaver study. J Hand Surg Eur Vol. 2016 Sep;41(7):683-7. doi: 10.1177/1753193416641319. Epub 2016 Apr 7. PMID 27056278
- [Result] Miller L, Crosbie J, Wajon A, Ada L. No difference between two types of exercise after proximal phalangeal fracture fixation: a randomised trial. J Physiother. 2016 Jan;62(1):12-9. doi: 10.1016/j.jphys.2015.11.006. Epub 2015 Dec 14. PMID 26699692
- [Derived] Zhang X, Yu Y, Shao X, Dhawan V, Du W. A randomized comparison of bone-cement K-wire fixation vs. plate fixation of shaft fractures of proximal phalanges. Phys Sportsmed. 2019 May;47(2):189-198. doi: 10.1080/00913847.2018.1546106. Epub 2018 Nov 14. PMID 30408421